CLINICAL TRIAL: NCT01638104
Title: ANX-042 Healthy Volunteer Dose Escalation Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Anexon, Incorporated (Industry); Celerion (Industry)
Responsible Party: Principal Investigator, Horng Chen, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ANX-042-C100
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- ANX-042: 0.001 mcg/kg/min (with low sodium diet) (Experimental): 0.001 dose unit equal to 1 millionth of a gram of an ANX-042 preparation / 1 kilogram of body mass administered / unit of time equal to 1 minute(mcg/kg/min), w/ diet restricted to 2.5 grams (gm) per day sodium (Na+) and 2.1 liters (L) fluid total daily intake
  Interventions: Drug: ANX-042
- ANX-042: 0.001 mcg/kg/min (Experimental): 0.001 mcg/kg/min ANX-042 with diet restricted to 4 gm per day Na+ and 3.6 L fluid total daily intake
  Interventions: Drug: ANX-042
- ANX-042: 0.003 mcg/kg/min (low sodium diet) (Experimental): 0.003 mcg/kg/min ANX-042 with diet restricted to 2.5 gm per day Na+ and 2.1 L fluid total daily intake
  Interventions: Drug: ANX-042
- ANX-042: 0.003 mcg/kg/min (Experimental): 0.003 mcg/kg/min ANX-042 with diet restricted to 4 gm per day Na+ and 3.6 L fluid total daily intake
  Interventions: Drug: ANX-042
- ANX-042: 0.0065 mcg/kg/min (low sodium diet) (Experimental): 0.0065 mcg/kg/min ANX-042 with diet restricted to 2.5 gm per day Na+ and 2.1 L fluid total daily intake
  Interventions: Drug: ANX-042
- ANX-042: 0.01 mcg/kg/min (low sodium diet) (Experimental): 0.01 mcg/kg/min ANX-042 with diet restricted to 2.5 gm per day Na+ and 2.1 L fluid total daily intake
  Interventions: Drug: ANX-042
- ANX-042: 0.01 mcg/kg/min (Experimental): 0.01 mcg/kg/min ANX-042 with diet restricted to 4 gm per day Na+ and 3.6 L fluid total daily intake
  Interventions: Drug: ANX-042
- ANX-042: 0.03 mcg/kg/min (Experimental): 0.03 mcg/kg/min ANX-042 with diet restricted to 4 gm per day Na+ and 3.6 L fluid total daily intake
  Interventions: Drug: ANX-042
- ANX-042: 0.1 mcg/kg/min (Experimental): 0.1 mcg/kg/min ANX-042 with diet restricted to 4 gm per day Na+ and 3.6 L fluid total daily intake
  Interventions: Drug: ANX-042
- ANX-042: 0.3 mcg/kg/min (Experimental): 0.3 mcg/kg/min ANX-042 with diet restricted to 4 gm per day Na+ and 3.6 L fluid total daily intake
  Interventions: Drug: ANX-042
- Placebo (low sodium diet) (Placebo Comparator): Placebo and diet restricted to 2.5 gm per day Na+ and 2.1 L fluid total daily intake
  Interventions: Drug: Placebo
- Placebo (Placebo Comparator): Placebo and diet restricted to 4 gm per day Na+ and 3.6 L fluid total daily intake
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ANX-042 — Reconstituted in Sterile Water for Injection, United States Pharmacopeia (USP) and administered by 12 hour continuous intravenous infusion with 5% dextrose in water (D5W), United States Pharmacopeia (USP)
  Arms: ANX-042: 0.001 mcg/kg/min; ANX-042: 0.001 mcg/kg/min (with low sodium diet); ANX-042: 0.003 mcg/kg/min; ANX-042: 0.003 mcg/kg/min (low sodium diet); ANX-042: 0.0065 mcg/kg/min (low sodium diet); ANX-042: 0.01 mcg/kg/min; ANX-042: 0.01 mcg/kg/min (low sodium diet); ANX-042: 0.03 mcg/kg/min; ANX-042: 0.1 mcg/kg/min; ANX-042: 0.3 mcg/kg/min
Drug: Placebo — Administered once by 12 hour continuous intravenous infusion with D5W (USP)
  Arms: Placebo; Placebo (low sodium diet)

SUMMARY:
The purpose of this study was to investigate the safety and tolerability of ANX-042 when administered by continuous intravenous (IV) infusion in healthy volunteers.

DETAILED DESCRIPTION:
Each participant received a total of two, approximately 12-hour continuous infusions of ANX-042 and one 12-hour continuous infusion of placebo, with a 36-hour washout period between treatments.

This study was conducted by Anexon, Inc. at Celerion, in Lincoln, Nebraska.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of non-reproductive potential (WNRP)

  * Men must be willing to use effective contraception and not donate sperm for up to 90 days after the final dose of study drug
  * Women must be of non-reproductive potential defined as a history of surgical sterilization or postmenopausal status (that is, greater than ( >) 50 years of age with >12 months amenorrhea while not using hormonal contraceptives or >50 years of age with 6-12 months of amenorrhea and follicle stimulating hormone (FSH) level >40 international unit/liter (IU/L)
* Good health status, physically active without cardio-respiratory limitations and minimal concomitant medications as determined by medical history and physical examination
* Able and willing to comply with study procedures, including controlled sodium (Na) intake and restriction of caffeine and tobacco product
* Have given written informed consent prior to the initiation of any study procedures

Exclusion Criteria:

* History of cardiovascular disease, unexplained syncope, postural tachycardia syndrome or frequent postural hypotension
* History or current evidence of respiratory, hepatic, renal, gastrointestinal, endocrine, hematological or neurological disorders that would constitute a risk when taking the study medication or interfere with the interpretation of data
* Clinically significantly abnormal clinical laboratory results (including Hepatitis B, Hepatitis C and Human Immunodeficiency Virus (HIV) serology) or physical examination results (confirmed by repeat measurement, if appropriate) that, in the opinion of the Investigator, would constitute a risk when taking the study medication or interfere with the interpretation of data
* Abnormal orthostatic Blood Pressure/Heart Rate (BP/HR) response at screening as defined by:

  * Systolic Blood Pressure (BP) decrease >20 millimeters of mercury (mmHg)
  * Diastolic BP decrease >10 mmHg, or
  * HR increase >25 beats per minute (bpm) and to a level above 100 bpm
* One or two supine values must be obtained between 8 and 10 minutes of supine rest. One or two upright values must be obtained between 3 and 5 minutes upright with the arm passively supported to maintain the brachial artery at heart level
* Abnormal 12-lead electrocardiogram (ECG) that interferes with proper measurement of QT-interval or, in the opinion of the Investigator, increases the risk of participating in the study
* Elevated BP (>140/90 mmHg) in any posture, confirmed by repeat measurement
* Current use (within 7 days of first dosing) or expected need for concomitant medications with hemodynamic effects including: non-steroidal anti-inflammatory drugs (NSAIDS), decongestants, BP medications, diuretics, monoamine oxidase inhibitors, norepinephrine uptake inhibitors (for example, attention-deficit disorder medications, anti-depressants) and erectile dysfunction medications. Medications with low likelihood of hemodynamic or renal effects are permitted (for example, acetaminophen, vitamins, stable thyroid hormone, gastritis therapies, antihistamines, topical medications, et cetera) after approval by the Investigator
* Evidence of current or recent use of known drugs of abuse and/or positive findings on urinary drug screening
* History of an average weekly alcohol intake that exceeds 21 units per week (1 unit equal to (=) 12 ounces (oz) or 360 milliliters (mL) of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits), or are unwilling to stop alcohol consumption for the duration of the study
* History of regular smoking of >5 cigarettes, cigars and/or pipe bowls of tobacco per day
* Known allergies to nesiritide (Natrecor)
* History of blood donation of >500 mL within one month, or plasma donation within 14 days, of first dosing
* Are currently enrolled in, or have completed or discontinued within the last 30 days from, a clinical trial involving an investigational product or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Are investigator site personnel directly affiliated with this study or their immediate family members. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted
* Are Lilly or Anexon employees or employees of any third-party organization (TPO) involved with the study that require exclusion of their employees

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with one or more drug-related adverse events (AEs) or any serious AEs | 0 to 4 weeks

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the plasma concentration-time curve (AUC) of ANX-042 | 0 to 24 hours post dose
Pharmacokinetics: Steady state plasma concentration of ANX-042 | 12 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Email: Anexon@Choruspharma.com, Study Director — Anexon, Incorporated
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No